CLINICAL TRIAL: NCT06960993
Title: Mosaic: RCT of a Digital Health Intervention for English- and Spanish-speaking Stem Cell Transplant Recipients
Brief Title: Mosaic Trial for Stem Cell Transplant Recipients
Acronym: Mosaic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Georgetown University (Other); Hackensack Meridian Health (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christine Rini, PhD, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00221336; R01CA292116 (NIH)
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Malignancy; Stem Cell Transplant; Bone Marrow Transplant; Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Website (Experimental): The intervention website pairs experiential information about transplant with (1) coordinated coping and stress management training and resources to support skill practice and (2) an educational component that includes educational content and links to well-established, vetted websites that provide broader, provider-reviewed information about the transplant process and links to psychosocial resources. Participants can toggle between English and Spanish content, and they will be able to use this website throughout their participation in the study.
  Interventions: Behavioral: Intervention website
- Enhanced Usual Care (Control) website (Active Comparator): The control website pairs (1) coordinated coping and stress management training and resources to support skill practice with (2) an educational component that includes educational content and links to well-established, vetted websites that provide broader, provider-reviewed information about the transplant process and links to psychosocial resources, using the same technology platform and look/feel as the intervention website.
  Participants can toggle between the English and Spanish versions of the website and they will be able to use this website throughout their participation in the study.
  Interventions: Behavioral: Enhanced Usual Care (Control) Website

INTERVENTIONS:
Behavioral: Intervention website — Website that includes experiential information, stress and coping resources, educational content, and links to trusted websites with additional educational content and links to psychosocial resources for transplant recipients and caregivers.
  Arms: Intervention Website
Behavioral: Enhanced Usual Care (Control) Website — Website that includes stress and coping resources, educational content, and links to trusted websites with additional educational content and links to psychosocial resources for transplant recipients and caregivers.
  Arms: Enhanced Usual Care (Control) website

SUMMARY:
The goal of this clinical trial is to learn if using an intervention website (Mosaic) improves selected patient-reported outcomes in adult blood cancer patients undergoing allogeneic or autologous stem cell transplant, compared to using an educational website (control group). Patients will be recruited prior to their scheduled transplant, then randomized to use one of these two study websites throughout the study. They will complete five assessments during the study: one before transplant (baseline) and four after transplant (2, 4, 6, and 8 month follow-ups).

The main questions this trial aims to answer are:

1. Compared to patients using the control group website, do patients using the intervention website report greater improvements in general psychological distress, cancer treatment-related distress, physical symptoms, and health-related quality of life?
2. Are these benefits at least partially explained by improvements in perceived preparedness, self-efficacy, and approach coping and/or reductions in avoidant coping and perceived stress?
3. Do some patients benefit more from using the intervention website than others? Specifically, we will examine whether patients' primary language (English/Spanish) and their initial psychological distress are related to the benefit they get from using the intervention website. We will also explore effects of sex, race, ethnicity, and transplant type.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a hematologic cancer according to medical records
* Scheduled for or preparing for scheduling of an allogeneic or autologous stem cell transplant at one of our study sites
* Aged 18 or older (no upper limit)
* English or Spanish Proficient
* Interested in using a website to learn about stem cell transplant
* Ability to understand and willingness to sign an informed consent document and comply with all study procedures

Exclusion Criteria:

* Currently participating in a behavioral intervention targeting distress, health-related quality of life, or symptoms
* Undergoing the first in a planned tandem stem cell transplant
* Unable to provide meaningful consent (severe cognitive impairment or language difficulties)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-06-12 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in general psychological distress | Baseline to 2 months post-transplant
  Improvement in general psychological measured with the PROMIS-57 Profile v2.1 emotional distress composite score. Raw scores are calculated and converted to T scores ranging from 0 to 100, with higher scores indicating more severe distress.

SECONDARY OUTCOMES:
Improvement in general psychological distress | Baseline to 4 months post-transplant
  Improvement in general psychological measured with the PROMIS-57 Profile v2.1 emotional distress composite score. Raw scores are calculated and converted to T scores ranging from 0 to 100, with higher scores indicating more severe distress.
Improvement in general psychological distress | Baseline to 6 months post-transplant
  Improvement in general psychological measured with the PROMIS-57 Profile v2.1 emotional distress composite score. Raw scores are calculated and converted to T scores ranging from 0 to 100, with higher scores indicating more severe distress.
Improvement in general psychological distress | Baseline to 8 months post-transplant
  Improvement in general psychological measured with the PROMIS-57 Profile v2.1 emotional distress composite score. Raw scores are calculated and converted to T scores ranging from 0 to 100, with higher scores indicating more severe distress.
Improvement in cancer treatment-related distress | Baseline to 2 months post-transplant
  Improvement in cancer treatment-related distress measured with the 23-item CTXD measure. The total score is calculated as the mean response across the items, yielding a score ranging from 0 to 3. Higher scores indicate greater distress.
Improvement in cancer treatment-related distress | Baseline to 4 months post-transplant
  Improvement in cancer treatment-related distress measured with the 23-item CTXD measure. The total score is calculated as the mean response across the items, yielding a score ranging from 0 to 3. Higher scores indicate greater distress.
Improvement in cancer treatment-related distress | Baseline to 6 months post-transplant
  Improvement in cancer treatment-related distress measured with the 23-item CTXD measure. The total score is calculated as the mean response across the items, yielding a score ranging from 0 to 3. Higher scores indicate greater distress.
Improvement in cancer treatment-related distress | Baseline to 8 months post-transplant
  Improvement in cancer treatment-related distress measured with the 23-item CTXD measure. The total score is calculated as the mean response across the items, yielding a score ranging from 0 to 3. Higher scores indicate greater distress.
Improvement in symptoms | Baseline to 2 months post-transplant
  Improvement in symptoms measured with the MDASI-Core. The measure's 13 core symptom items assess the severity of symptoms on a 0-10 numerical rating scale from 0 (not present) to 10 (as bad as you can imagine). These ratings are averaged into symptom severity score ranging from 0 to 10, with higher scores indicating more severe symptoms.
Improvement in symptoms | Baseline to 4 months post-transplant
  Improvement in symptoms measured with the MDASI-Core. The measure's 13 core symptom items assess the severity of symptoms on a 0-10 numerical rating scale from 0 (not present) to 10 (as bad as you can imagine). These ratings are averaged into symptom severity score ranging from 0 to 10, with higher scores indicating more severe symptoms.
Improvement in symptoms | Baseline to 6 months post-transplant
  Improvement in symptoms measured with the MDASI-Core. The measure's 13 core symptom items assess the severity of symptoms on a 0-10 numerical rating scale from 0 (not present) to 10 (as bad as you can imagine). These ratings are averaged into symptom severity score ranging from 0 to 10, with higher scores indicating more severe symptoms.
Improvement in symptoms | Baseline to 8 months post-transplant
  Improvement in symptoms measured with the MDASI-Core. The measure's 13 core symptom items assess the severity of symptoms on a 0-10 numerical rating scale from 0 (not present) to 10 (as bad as you can imagine). These ratings are averaged into symptom severity score ranging from 0 to 10, with higher scores indicating more severe symptoms.
Improvement in health-related quality of life | Baseline to 2 months post-transplant
  Improvement in health-related quality of life measured with the PROMIS Global-10 scale V1.2. Final scores are created by summing responses to each of the 10 items, then converting the raw score into two summary T-scores, each ranging from 0-100: one for Global Physical Health and one for Global Mental Health. Higher scores indicate better quality of life in the given domain.
Improvement in health-related quality of life | Baseline to 4 months post-transplant
  Improvement in health-related quality of life measured with the PROMIS Global-10 scale V1.2. Final scores are created by summing responses to each of the 10 items, then converting the raw score into two summary T-scores, each ranging from 0-100: one for Global Physical Health and one for Global Mental Health. Higher scores indicate better quality of life in the given domain.
Improvement in health-related quality of life | Baseline to 6 months post-transplant
  Improvement in health-related quality of life measured with the PROMIS Global-10 scale V1.2. Final scores are created by summing responses to each of the 10 items, then converting the raw score into two summary T-scores, each ranging from 0-100: one for Global Physical Health and one for Global Mental Health. Higher scores indicate better quality of life in the given domain.
Improvement in health-related quality of life | Baseline to 8 months post-transplant
  Improvement in health-related quality of life measured with the PROMIS Global-10 scale V1.2. Final scores are created by summing responses to each of the 10 items, then converting the raw score into two summary T-scores, each ranging from 0-100: one for Global Physical Health and one for Global Mental Health. Higher scores indicate better quality of life in the given domain.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Georgetown University School of Medicine, Washington D.C., District of Columbia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Hackensack Meridian Health, Nutley, New Jersey

IPD SHARING:
Plan to Share IPD: No
We will not be sharing IPD